CLINICAL TRIAL: NCT01398371
Title: A Randomised, Blinded, Placebo Controlled Trial to Assess the Effect of Digoxin Withdrawal in Stable Heart Failure Patients Receiving Optimal Background Therapy
Brief Title: Digoxin Withdrawal in Stable Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Dr Ingrid Hopper, The Alfred
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 257/11; Pending (Other Grant/Funding Number: Pending)
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
Keywords: Heart failure; Digoxin withdrawal
MeSH Terms: conditions — Heart Failure | interventions — Digoxin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stable digoxin therapy (Active Comparator): Participants need to have been receiving digoxin therapy for at least 3 months at a dose that results in digoxin plasma levels of 0.4-0.8 on 2 consecutive blood tests (at least 1 weeks apart) prior to randomisation. The dose of digoxin must remain stable for at least 2 weeks prior to randomisation.
  Interventions: Drug: Digoxin
- Digoxin withdrawal (Experimental): Participants will receive a placebo for 4 weeks.
  Interventions: Drug: Withdrawal of digoxin

INTERVENTIONS:
Drug: Withdrawal of digoxin — Participants currently receiving digoxin for heart failure will have their digoxin stopped for 12 weeks.
  Arms: Digoxin withdrawal
Drug: Digoxin — Stable digoxin therapy which produces a digoxin plasma level of 0.4-0.8.
  Arms: Stable digoxin therapy

SUMMARY:
Heart failure is a chronic condition in which the heart fails to function as a pump to move blood around the body. This sets up a complex physiologic response to compensate, which include activation of many hormonal mechanisms which result in fluid accumulation.

In recent years, medications to block the hormonal response to heart failure are given as standard drugs, and these include ACE inhibitors, and beta blockers. Mortality is reduced with these medications, as well as symptoms improved.

Medications that were traditionally used in heart failure include diuretics, which cause fluid loss, and digoxin, which causes the heart to pump harder. These medications were introduced before clinical trials as we know them now were run. Since the introduction of ACE inhibitors and beta blockers, it is not clear whether there is still a role for digoxin.

In this study, we plan to withdraw digoxin from patients with stable heart failure in normal rhythm, taking stable doses of ACE inhibitors and beta blockers, in a closely monitored environment and watch for the effect of this on heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years
2. In sinus rhythm at the time of randomisation
3. Have a LVEF <0.45 and a left ventricular end-diastolic dimension >60 mm or >34 mm/m2
4. Are receiving ACE inhibitor, β-blocker and diuretic therapy at the optimal doses.
5. Has been receiving digoxin therapy for at least 3 months at a dose that results in digoxin plasma levels of 0.4-0.8 on 2 consecutive blood tests (at least 1 weeks apart) prior to randomisation. The dose of digoxin must remain stable for at least 2 weeks prior to randomisation.
6. Documented, stable heart failure. Must have at least 1 of the following:

   * Hospitalised with a discharge diagnosed of heart failure in the last 6 months
   * Evidence of pulmonary congestion on chest X-ray
   * Evidence of heart failure on echocardiogram
   * Evidence of heart failure on ECG
7. Willing and able to provide informed consent

Exclusion Criteria:

1. Systolic BP >160mmHg or <90mmHg
2. Diastolic BP >95mmHg
3. Uncorrected primary valvular disease
4. Active myocarditis
5. Obstructive or restrictive Cardiomyopathy
6. Exercise capacity limited by other factors not including dyspnoea
7. Myocardial infarction within the previous 6 months
8. Stroke within the previous 12 months
9. Hospitalisation within one month of randomisation
10. A history of supraventricular arrhythmia or sustained ventricular arrhythmia
11. Claudication
12. Severe primary pulmonary (VC <1.5L), renal or hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
NYHA Heart Failure class | after 12 wks of treatment

SECONDARY OUTCOMES:
6 minute walk test | after 12 wks of treatment
Quality of Life | After 12 weeks of treatment
  Standard questionnaires will be used
Change in BNP | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS, FRACP, PhD, Principal Investigator — Alfred Hospital / Monash University
Locations (1):
- Clinical Pharmacology, Alfred Hospital, Melbourne, Victoria, Australia